CLINICAL TRIAL: NCT01030380
Title: Determination of the Efficacy of Slendertone® Face to Tone the Muscles of the Face and Reduce the Signs of Facial Aging
Acronym: Face
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Dr. Michael Hennessy, Principal Investigator, Neurologist
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMR-09-2009
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Facial Muscle Toning
Keywords: Facial toning; Facial lift; Improve facial complexion; Improve facial tone; Improve radiance of the face; Reduce signs of facial aging; firming, lift, tone face

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slendertone Face NMES (Experimental): Slendertone Face 20 minutes/day, 5 days/week for 12 weeks.
  Interventions: Device: Slendertone Face
- Control Group: No NMES (No Intervention): Control Group: No NMES over the course of 12 weeks.

INTERVENTIONS:
Device: Slendertone Face — Slendertone Face 20 minutes/day, 5 days/week for 12 weeks.
  Other Names: Slendertone Face, Type 371; Class II, Powered Muscle Stimulator
  Arms: Slendertone Face NMES

SUMMARY:
The purpose of this study was to determine the efficacy of Slendertone® Face™, to tone the muscles of the face and reduce the signs of facial aging among the following characteristics: radiance, tone, lift, firmness and complexion, following a 12-week programme of facial muscle toning. Slendertone® Face is a neuromuscular electrical stimulation (NMES) device which features a headset unit designed for application to the face for facial toning. The purpose of the headset is to locate and support a pair of stimulation electrodes on each side of the face, over the facial nerve just anterior to the ear.

DETAILED DESCRIPTION:
The trial was planned with 100 healthy female volunteers between 25 and 55 years of age.

Treated group: Face device 20 minutes per day, 5 days per week for 12 weeks.

Control group: No NMES.

Both Groups: No changes to usual beauty routine, or use of beauty products with an anti-aging claim, or changes to usual diet or exercise habits over the course of the 12 week study period.

Assessments:

Ultrasound measurements of the zygomaticus major muscle were planned at Baseline, and at the end of Weeks 6 and 12.

Psychometric questionnaires at Baseline, end of Weeks 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (by their own report) female participants aged between 35 and 55
* Visual signs of aging of the face
* Able and willing to complete all study assessments and to be followed for the full course of the study.
* Able to read, write and follow instructions in English.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnant women (or pregnancy within last 3 months).
* Inadequate precaution or procedure to prevent pregnancy (women of child- bearing potential only).
* Individuals who have any implanted medical devices (pacemaker, pump, catheter, etc.)
* Current or history of a medical condition that would contraindicate treatment with the product, such as epilepsy, hernia, abdominal ulcer, diabetes, or other conditions which, in the opinion of the Investigator, would place the participant at risk.
* A current skin disease of any type at the test site (e.g. acne, eczema, psoriasis, burns, abrasions, etc.)
* Heavy alcohol consumption in the opinion of the investigator.
* A fever in the last 12 hours prior to the first application of the test device.
* History of heart disease.
* History of stroke.
* History of malignant disease.
* Insulin dependent diabetes.
* Concurrent medication likely to affect the response to the test article or confuse the results of the study (e.g. routine high dose use of any drugs that may artificially affect skin tone).
* Individuals who are currently participating in any other clinical. investigation, or who have participated in a study with the same indication within 1 year.
* Principal investigator for this study, or member of study staff.
* Individuals who have had facial surgery.
* Individuals who use BOTOX. (The latter two exclusions were applied because of the possibility of an altered anatomical or physiological background which may have interfered with the effectiveness of the treatment).

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Ultrasound measurements of the zygomaticus major muscle | Baseline; End of Week 6; End of Week 12
Increased psychometric assessments of improvements among the characteristics of facial appearance: firming; tone; lift; radiance and complexion | Baseline; End of Week 6 and End of Week 12

SECONDARY OUTCOMES:
Ease of Use and Overall Acceptance of the Slendertone Face device | End of Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hennessy, M.D., Principal Investigator — Chief of Neurology, Galway University Hospital
Locations (1):
- Bio-Medical Research, Ltd., Galway, County Galway, Ireland

REFERENCES:
- [Background] Coleman SR, Grover R. The anatomy of the aging face: volume loss and changes in 3-dimensional topography. Aesthet Surg J. 2006 Jan-Feb;26(1S):S4-9. doi: 10.1016/j.asj.2005.09.012. PMID 19338976
- [Background] Rexbye H, Petersen I, Johansens M, Klitkou L, Jeune B, Christensen K. Influence of environmental factors on facial ageing. Age Ageing. 2006 Mar;35(2):110-5. doi: 10.1093/ageing/afj031. Epub 2006 Jan 11. PMID 16407433
- [Background] Roubenoff R. Sarcopenia and its implications for the elderly. Eur J Clin Nutr. 2000 Jun;54 Suppl 3:S40-7. doi: 10.1038/sj.ejcn.1601024. PMID 11041074
- [Background] Branchet MC, Boisnic S, Frances C, Robert AM. Skin thickness changes in normal aging skin. Gerontology. 1990;36(1):28-35. doi: 10.1159/000213172. PMID 2384222
- [Background] Zimbler MS, Kokoska MS, Thomas JR. Anatomy and pathophysiology of facial aging. Facial Plast Surg Clin North Am. 2001 May;9(2):179-87, vii. PMID 11457684
- [Background] McMiken DF, Todd-Smith M, Thompson C. Strengthening of human quadriceps muscles by cutaneous electrical stimulation. Scand J Rehabil Med. 1983;15(1):25-8. PMID 6828830
- [Background] Charette SL, McEvoy L, Pyka G, Snow-Harter C, Guido D, Wiswell RA, Marcus R. Muscle hypertrophy response to resistance training in older women. J Appl Physiol (1985). 1991 May;70(5):1912-6. doi: 10.1152/jappl.1991.70.5.1912. PMID 1864770
- [Background] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Background] Porcari JP, Miller J, Cornwell K, Foster C, Gibson M, McLean K, Kernozek T. The effects of neuromuscular electrical stimulation training on abdominal strength, endurance, and selected anthropometric measures. J Sports Sci Med. 2005 Mar 1;4(1):66-75. eCollection 2005 Mar 1. PMID 24431963
- [Background] Quittan M, Wiesinger GF, Sturm B, Puig S, Mayr W, Sochor A, Paternostro T, Resch KL, Pacher R, Fialka-Moser V. Improvement of thigh muscles by neuromuscular electrical stimulation in patients with refractory heart failure: a single-blind, randomized, controlled trial. Am J Phys Med Rehabil. 2001 Mar;80(3):206-14; quiz 215-6, 224. doi: 10.1097/00002060-200103000-00011. PMID 11237275
- [Background] Vanderthommen M, Depresseux JC, Dauchat L, Degueldre C, Croisier JL, Crielaard JM. Spatial distribution of blood flow in electrically stimulated human muscle: a positron emission tomography study. Muscle Nerve. 2000 Apr;23(4):482-9. doi: 10.1002/(sici)1097-4598(200004)23:43.0.co;2-i. PMID 10716757